CLINICAL TRIAL: NCT05227677
Title: Value of Glycated Albumin in Intervention of Glycemic Control in Patients With Type 2 Diabetes: A Multicenter, Randomized Controlled Clinical Study
Brief Title: Value of Glycated Albumin in Intervention of Glycemic Control in Chinese Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAID1
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; glycated albumin; intervention; anti-diabetic regimens; Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A total of 200 patients with newly diagnosed T2DM will be 1:1 randomly assigned to two groups: intervention group (GA) and control group (NC). After testing baseline metabolic indexes including A1c, all the patients will be treated with antidiabetic therapy according to guideline for prevention and treatment of type 2 diabetes in China (2020) and followed up for 12 weeks. The GA concentration will be measured at 4-week intervals. In GA group, the anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks. In NC group, investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment. At the end of 12 weeks, A1c and other metabolic indexes will be measured again. All the anti-diabetic drugs are permitted in this study except sulfonylureas, glinides, insulin and insulin analogues.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA guided anti-diabetic therapy adjustment (Experimental): The GA values will be measured at 4-week intervals and the anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks.
  Interventions: Other: GA guided anti-diabetic therapy adjustment
- current guidelines to adjust treatment (Active Comparator): The GA values will be measured at 4-week intervals，but investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment.
  Interventions: Other: current guidelines to adjust treatment

INTERVENTIONS:
Other: GA guided anti-diabetic therapy adjustment — The GA values will be measured at 4-week intervals in both groups. The anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks.
  Arms: GA guided anti-diabetic therapy adjustment
Other: current guidelines to adjust treatment — The GA values will be measured at 4-week intervals. Investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment.
  Arms: current guidelines to adjust treatment

SUMMARY:
HbA1c is widely used as the gold standard for evaluating glycemic control. However, in patients who need adjusting hypoglycemic regimen, A1c was not a sensitive marker. In comparison, serum GA level can reflect the average blood glucose level in the last 2~3 weeks of diabetes.

Therefore, investigators undertake this study to determine whether knowledge of GA values and adjusting anti-diabetic regimens according to GA values will result in improved glycemic control in newly diagnosed type 2 diabetes mellitus (T2DM).

This multicenter randomized controlled clinical study will be conducted in 10 hospitals in China. A total of 200 patients with newly diagnosed T2DM will be 1:1 randomly assigned to two groups: intervention group (GA) and control group (NC). In GA group, the anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks. In NC group, investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment. At 12-week of follow-up，investigators compare the achievement rate of HbA1c(<7%) between the two groups.

DETAILED DESCRIPTION:
At present, glycosylated hemoglobin (HbA1c) is widely used as the gold standard for evaluating glycemic control. However, as a marker of average blood glucose level, HbA1c has some limitations. HbA1c is affected by many conditions, such as hemolytic anemia, recent blood loss or blood transfusion, chronic renal failure, the use of erythropoietin or other drugs affecting hematopoiesis, and the presence of variant hemoglobin. In addition, HbA1c represents the average blood glucose level in the last 2-3 months, in patients who need adjusting hypoglycemic regimen, A1c was not a sensitive marker. Therefore, finding clinical markers that can timely guide the adjustment and evaluate therapeutic effects is an urgent demand for individualized treatment of diabetes.

Glycated albumin (GA) has been available in clinic for sixteen years, yet the clinical value of routine measurements of GA in the care of diabetic patients is still uncertain. Previous studies have shown that the GA half-life is 17-19 days, so the serum GA level can reflect the average blood glucose level and the recent blood glucose changes and the extent of the changes in the last 2~3 weeks of diabetes, and is not affected by age, gender, diet, drugs and glycemic fluctuation. A recent short-term study found that in newly diagnosed type 2 diabetic patients with initial therapy and in patients with type 2 diabetes and unsatisfactory glucose control and need intensifying treatment, changes in GA could predict changes in HbA1c levels after 3 months. Therefore, investigators undertake this study to determine whether knowledge of GA values and adjusting anti-diabetic regimens according to GA values will result in improved glycemic control in newly diagnosed type 2 diabetes mellitus (T2DM).

This multicenter randomized controlled clinical study will be conducted in 10 hospitals in China. A total of 200 patients with newly diagnosed T2DM will be 1:1 randomly assigned to two groups: intervention group (GA) and control group (NC). In this study, the clinical related indexes such as GA, fasting blood glucose, HbA1c, fasting C-peptide, fasting insulin, liver and kidney function, blood routine, blood uric acid and blood lipid were measured at baseline. The GA serum was frozen and not used as the basis for initial treatment. All the patients will be treated with antidiabetic therapy according to guideline for prevention and treatment of type 2 diabetes in China (2020) and followed up for 12 weeks. The GA concentration will be measured at 4-week intervals. In GA group, the anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks. In NC group, investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment. At the end of 12 weeks, A1c and other metabolic indexes will be measured again. All the anti-diabetic drugs are permitted in this study except sulfonylureas, glinides, insulin and insulin analogues.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years of age
* newly diagnosed T2DM or duration of T2DM less than 1 year and without anti-diabetic medications for 3 months prior to screening
* HbA1c ≥7.5% and <10.5%

Exclusion Criteria:

* Requiring treatment of proliferative retinopathy, maculopathy, painful diabetic neuropathy, diabetic foot, diabetic ketoacidosis, or hyperglycemic hyperosmolar status in recent 3 months prior to screening.
* The following history or conditions in recent 6 months prior to screening: (i) decompensated cardiac insufficiency (NYHA class III or IV); (ii)myocardial infarction, coronary artery bypass grafting or coronary stent implantation; (iii) uncontrolled severe arrhythmia and is not suitable to participate in this study evaluated by the investigator; (iv) hemorrhagic stroke or ischemic stroke and is not suitable to participate in this study evaluated by the investigator.
* Laboratory indicators meet one of the following criteria: (i) alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3× upper limit of normal(ULN); (ii) total bilirubin > 2× ULN; (iii) hemoglobin <100g/L; (iv)total protein <60g/L; (v)albumin <30g/L; (vi) glomerular filtration rate(eGFR)<60 ml min-1 per 1.73 m2.
* Thalassemia, hemolytic anemia and other diseases that may cause erythrocyte instability and affect the measurement of HbA1c.
* Uncontrolled thyroid dysfunction.
* Systemic corticosteroids treatment in recent 1 month prior to screening (exception of inhalation or local external treatment).
* Pregnancy or lactating.
* Two or more episodes of severe hypoglycemia in recent 1 year prior to screening.
* Patient who need to initiate treatment with sulfonylureas, glinides, insulin or insulin analogues evaluated by the investigators.
* Patient is being treated with calcium dobesilate or has a disease requiring calcium dobesilate treatment, or may be treated with calcium dobesilate in the near future evaluated by the investigators.
* Patients considered unsuitable for observation by investigators.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Professor, Principal Investigator — Peking University People's Hospital
Locations (7):
- China (7):
  - The third people's hospital of DATONG, Datong, Shanxi
  - Beijing Haidian Hospital, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - Beijing Shijingshan Hospital, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Civil Aviation General Hospital, Beijing
  - Peking University People's Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ren Q, Ji LN, Lu JM, Li YF, Li QM, Lin SS, Lv XF, Wang L, Xu Y, Guo XH, Guo QY, Ma L, Du J, Chen YL, Zhao CL, Zhang QL, She QM, Jiao XM, Lu MH, Sun XM, Gao Y, Zhang J. Search for clinical predictors of good glycemic control in patients starting or intensifying oral hypoglycemic pharmacological therapy: A multicenter prospective cohort study. J Diabetes Complications. 2020 Feb;34(2):107464. doi: 10.1016/j.jdiacomp.2019.107464. Epub 2019 Oct 20. PMID 31771933
- [Background] Lu JM, Ji LN, Li YF, Li QM, Lin SS, Lv XF, Wang L, Xu Y, Guo XH, Guo QY, Ma L, Du J, Chen YL, Zhao CL, Zhang QL, She QM, Jiao XM, Lu MH, Pan RQ, Gao Y. Glycated albumin is superior to glycated hemoglobin for glycemic control assessment at an early stage of diabetes treatment: A multicenter, prospective study. J Diabetes Complications. 2016 Nov-Dec;30(8):1609-1613. doi: 10.1016/j.jdiacomp.2016.07.007. Epub 2016 Jul 16. PMID 27496253
- See also: Articles related to clinical trials — https://www.healio.com/news/endocrinology/20191025/glycated-albumin-good-predictor-when-assessing-glucose-management

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 207 participants, 11 were excluded for reasons such as not meeting criteria for newly diagnosed type 2 diabetes, unsuitable for observation, age requirements, protocol violation, and mistaken inclusion. 196 participants were successfully screened, and 200 were randomly assigned to the study. Four participants violated criteria but were still included. The study groups consisted of 98 in the intervention group and 102 in the control group.
Groups:
- GA guided anti-diabetic therapy adjustment: The Glycated ALbumin (GA) value will be measured at 4-week intervals and the anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks.
  GA guided anti-diabetic therapy adjustment: The GA concentration will be measured at 4-week intervals in both groups. The anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks.
- current guidelines to adjust treatment: The GA concentration will be measured at 4-week intervals，but investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment.
  current guidelines to adjust treatment: The GA concentration will be measured at 4-week intervals. Investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment.
Period: Overall Study
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Started | 98 | 102
Completed | 86 | 93
Not Completed | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- GA Guided Anti-diabetic Therapy Adjustment: The Glycated Albumin (GA) value will be measured at 4-week intervals and the anti-diabetic treatment regimen will be strengthened when GA values is higher than 16% at 4 weeks.
- Current Guidelines to Adjust Treatment: The GA value will be measured at 4-week intervals，but investigators will be not aware of the GA value and rely on the current guidelines to adjust treatment.
- Total: Total of all reporting groups
Arm/Group | GA Guided Anti-diabetic Therapy Adjustment | Current Guidelines to Adjust Treatment | Total
Number analyzed (Participants) | 98 | 101 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (10.76) | 50.7 (10.65) | 50.0 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 36 | 68
  Male | 66 | 65 | 131
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 98 | 101 | 199
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 28.2 (3.5) | 27.7 (4.5) | 27.9 (4.0)
Waist circumference [Mean (Standard Deviation); unit: cm] | 97.0 (8.4) | 94.7 (11.2) | 95.9 (10.0)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 135 (17) | 133 (13) | 134 (16)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 86 (11) | 85 (11) | 85 (11)
Participants with Hyperlipidemia [Count of Participants; unit: Participants] | 57 | 55 | 112
Participants with Hypertension [Count of Participants; unit: Participants] | 36 | 41 | 77
Fasting Blood Glucose [Mean (Standard Deviation); unit: mmol/L] | 9.93 (1.93) | 9.31 (1.83) | 9.63 (1.89)
HbA1c [Mean (Standard Deviation); unit: %] | 8.9 (0.9) | 8.7 (0.8) | 8.8 (8.9)
Glycated Albumin [Mean (Standard Deviation); unit: %] | 22.5 (4.1) | 21.9 (3.5) | 22.2 (3.8)
Fasting serum insulin [Median (Inter-Quartile Range); unit: μU/mL] | 11.73 [7.99 to 17.40] | 11.55 [8.32 to 18.50] | 11.70 [7.99 to 18.36]
Fasting serum C peptide [Median (Inter-Quartile Range); unit: ng/mL] | 2.91 [2.26 to 3.71] | 2.88 [2.16 to 3.51] | 2.89 [2.17 to 3.71]
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) [Median (Inter-Quartile Range); unit: FINS(μIU)×FPG(mmol/L)/22.5] | 5.30 [3.50 to 7.40] | 4.80 [3.30 to 7.90] | 5.15 [3.35 to 7.52]
HOMA-β [Median (Inter-Quartile Range); unit: 20×FINS(μIU/mL)/(FPG(mmol/L)-3.5)] | 37.6 [24.5 to 63.6] | 43.7 [25.9 to 75.6] | 40.0 [25.6 to 67.3]
Leucocyte [Mean (Standard Deviation); unit: cells*10^9/L] | 6.65 (1.46) | 7.18 (1.97) | 6.92 (1.76)
Erythrocyte [Mean (Standard Deviation); unit: cells*10^9/L] | 5.02 (0.44) | 5.06 (0.52) | 5.05 (0.47)
Platelet [Mean (Standard Deviation); unit: cells*10^9/L] | 245 (63.4) | 241 (59.0) | 242.8 (61.2)
Hemoglobin [Mean (Standard Deviation); unit: g/L] | 153.5 (16.02) | 153.8 (14.26) | 153.8 (15.00)
Alanine Aminotransferase (ALT) [Median (Inter-Quartile Range); unit: U/L] | 33.3 [21.2 to 49.0] | 35.4 [22.4 to 50.1] | 34.9 [21.3 to 50.0]
Serum Creatinine [Mean (Standard Deviation); unit: μmol/L] | 66.5 (14.1) | 65.2 (15.0) | 65.8 (14.6)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m2] | 106.3 (18.1) | 106.0 (18.3) | 106.3 (18.0)
Serum uric acid [Median (Inter-Quartile Range); unit: μmol/L] | 348.4 [277.0 to 398.1] | 323.0 [281.0 to 370.0] | 338.5 [280.8 to 389.8]
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.36 (1.11) | 5.17 (0.99) | 5.26 (1.02)
triglyceride [Median (Inter-Quartile Range); unit: mmol/L] | 2.08 [1.48 to 2.85] | 1.92 [1.38 to 3.15] | 2.00 [1.41 to 3.01]
HDL-C [Mean (Standard Deviation); unit: mmol/L] | 1.14 (0.25) | 1.18 (0.26) | 1.16 (0.25)
LDL-C [Mean (Standard Deviation); unit: mmol/L] | 3.43 (1.00) | 3.25 (0.86) | 3.34 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: The Achievement Rate of HbA1c (<7%)
Description: To compare the achievement rate of HbA1c(<7%) between the two groups at 12-week of follow-up.
Time Frame: 12 weeks
Population: Analysis dataset included two sets. Full analysis set (FAS) was defined as participants who were randomized, met the study inclusion criteria, and had baseline measurements of the primary efficacy endpoint. Per protocol set (PPS) was defined as subjects with good compliance in FAS and no significant protocol deviations that affect the primary efficacy evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- GA guided anti-diabetic therapy adjustment: The GA concentration will be measured at 4-week intervals and the anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks.
  GA guided anti-diabetic therapy adjustment: The GA concentration will be measured at 4-week intervals in both groups. The anti-diabetic treatment regimen will be strengthened when GA value is higher than 16% at 4 weeks.
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 98 | 101
Participants
  FAS analysis | 63 | 65
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | 58 | 64
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; Test type: Superiority — FAS analysis; p = 0.9917, Chi-squared — The threshold for statical significance was p=0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.6555, Chi-squared

2. Secondary Outcome: The Achievement Rate of HbA1c(<6.5%)
Description: To compare the achievement rate of HbA1c(<6.5%) between the two groups at 12-week of follow-up.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 98 | 101
Participants
  FAS analysis | 35 | 24
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | 32 | 23
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0649, Chi-squared — The threshold for statical significance was p=0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0342, Chi-squared

3. Secondary Outcome: The Achievement Rate of HbA1c (<6%)
Description: To compare the achievement rate of HbA1c(<6%) between the two groups at 12-week of follow-up.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 98 | 101
Participants
  FAS analysis | 13 | 8
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | 13 | 7
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS Analysis; Test type: Superiority; p = 0.2199, Chi-squared — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority — The threshold for statistical significance was p =0.05; p = 0.0769, Chi-squared

4. Secondary Outcome: Change in HbA1c Levels
Description: To compare the change of HbA1c levels between the two groups after 12-week of follow-up.
Time Frame: 12 weeks
Population: At V5, HbA1c measurements were unavailable for 12 participants in the GA intervention group and 8 participants in the control group. Consequently, the FAS analysis of HbA1c changes was conducted using data from 86 participants in the GA intervention group and 93 participants in the control group.
Measure: Median (Inter-Quartile Range); unit: percentage of HbA1c
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
percentage of HbA1c
  FAS analysis | -2.3 [-2.9 to -1.5] | -1.7 [-2.5 to -1.2]
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -2.3 [-3.0 to -1.5] | -1.7 [-2.5 to -1.2]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0200, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0147, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rate of Change in HbA1c Levels
Description: To compare the rate of change in HbA1c measurements between the two groups after 12-week of follow-up.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
Percent change
  FAS analysis | -24.794 (9.8781) | -21.574 (9.2575)
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -24.971 (10.0353) | -21.474 (9.0570)
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0256, t-test, 2 sided — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0181, t-test, 2 sided — The threshold for statistical significance was p =0.05

6. Secondary Outcome: Rate of Hypoglycemic Events
Description: To compare the rate of hypoglycemic events between the two groups
Time Frame: at visit 3(4 weeks) and visit 4(8 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 98 | 101
Participants
  FAS analysis at V3 | 1 | 1
  FAS analysis at V4 | 2 | 1
  PPS analysis at V3: number analyzed (Participants) | 79 | 91
  PPS analysis at V3 | 1 | 1
  PPS analysis at V4: number analyzed (Participants) | 79 | 91
  PPS analysis at V4 | 2 | 1
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; At Visit3 (FAS); Test type: Equivalence — Compare the percentage of hypoglycemia in each group and whether the percentage of hypoglycemia is equivalent between the GA guided therapy group and the Standard therapy group; p > 0.999, Fisher Exact — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; At Visit 4 (FAS); Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.6175, Fisher Exact — The threshold for statistical significance was p =0.05
Statistical Analysis 3: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; At Visit 3 (PPS); Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p > 0.999, Fisher Exact — The threshold for statistical significance was p =0.05
Statistical Analysis 4: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; At Visit4 (PPS); Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.5979, Fisher Exact — The threshold for statistical significance was p =0.05

7. Secondary Outcome: Change in HOMA-β Levels
Description: To compare the change in HOMA-β levels between the two groups after 12-week of follow-up.
Time Frame: 12 weeks
Population: At V5, HOMA-β data were missing for 12 participants in the GA intervention group (GA) and 10 in the control group, resulting in FAS analysis using 86 GA and 91 control participants. In the PPS group, data were missing for 0 in GA and 2 in control, so PPS analysis included 79 GA and 89 control participants.
Measure: Median (Inter-Quartile Range); unit: percentage of beta cell function
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 91
percentage of beta cell function
  FAS analysis | 33.60 [15.70 to 59.00] | 21.50 [9.50 to 47.00]
  PPS analysis: number analyzed (Participants) | 79 | 89
  PPS analysis | 33.70 [15.70 to 59.30] | 21.50 [10.40 to 43.80]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0404, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0330, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Percent Change in HOMA-β Levels
Description: To compare the rate in change of HOMA-β levels between the two groups after 12-week of follow-up.
Time Frame: 12 weeks
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Percent change in HOMA-β
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 91
Percent change in HOMA-β
  FAS analysis | 89.10 [33.30 to 184.00] | 66.30 [23.20 to 121.50]
  PPS analysis: number analyzed (Participants) | 79 | 89
  PPS analysis | 90.30 [33.30 to 207.40] | 66.30 [24.00 to 116.00]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0408, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0322, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

9. Secondary Outcome: Change in HOMA-IR Levels
Description: To compare the change in HOMA-IR between two groups after 12 weeks of follow-up.
  The HOMA-IR (Homeostasis Model Assessment of Insulin Resistance) index is a widely used surrogate marker for assessing insulin resistance. It is calculated as:
  HOMA-IR = (Fasting Insulin [μU/mL] × Fasting Glucose [mg/dL]) / 405
  Interpretation:
  Lower HOMA-IR values indicate better insulin sensitivity. Higher HOMA-IR values suggest increased insulin resistance.
  Typical Reference Ranges:
  1.0-1.9: Normal range 2.0-2.9: Early insulin resistance
  ≥3.0: Significant insulin resistance
  Note: These ranges may vary depending on population characteristics and laboratory standards. There is no universally defined theoretical minimum or maximum value. Clinical thresholds such as ≥2.5 or ≥3.0 are commonly used to indicate insulin resistance in adults.
Time Frame: 12 weeks
Population: At V5, HOMA-IR data were missing for 12 participants in the GA intervention group (GA) and 10 in the control group, resulting in FAS analysis using 86 GA and 91 control participants. In the PPS group, data were missing for 0 in GA and 2 in control, so PPS analysis included 79 GA and 89 control participants.
Measure: Median (Inter-Quartile Range); unit: index
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 91
index
  FAS analysis | -2.10 [-3.30 to -0.50] | -1.10 [-2.60 to 0.20]
  PPS analysis: number analyzed (Participants) | 79 | 89
  PPS analysis | -2.30 [-3.30 to -0.60] | -1.10 [-2.60 to 0.10]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0303, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0264, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

10. Secondary Outcome: Percent Change in HOMA-IR Levels
Description: To compare the rate of change in HOMA-IR levels between the two groups after 12-week of follow-up.
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Percent Change in HOMA-IR
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 91
Percent Change in HOMA-IR
  FAS analysis | -42.35 [-57.40 to -14.30] | -27.50 [-51.40 to 5.60]
  PPS analysis: number analyzed (Participants) | 79 | 89
  PPS analysis | -43.80 [-57.40 to -20.80] | -30.00 [-51.40 to 4.3]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0374, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0313, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

11. Secondary Outcome: Change in Weight
Description: To compare the change in weight between two groups after 12 weeks of follow-up.
Time Frame: 12 weeks
Population: At V5, Weight data were missing for 12 participants in the GA intervention group (GA) and 8 in the control group, resulting in FAS analysis using 86 GA and 93 control participants. In the PPS group, no data were missing for in GA and in control, so PPS analysis included 79 GA and 91 control participants.
Measure: Median (Inter-Quartile Range); unit: Weight Change(kg)
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
Weight Change(kg)
  FAS analysis | -2.45 [-5.00 to -0.700] | -1.50 [-3.20 to 0.00]
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -2.40 [-5.10 to -0.70] | -1.50 [-3.30 to 0.00]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0086, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0156, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Percent Change in Weight
Description: To compare the rate of change in weight between the two groups at 12-week of follow-up.
Time Frame: 12weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Percent Change in Weight
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
Percent Change in Weight
  FAS analysis | -2.940 [-6.520 to -0.720] | -1.670 [-4.410 to 0.000]
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -2.930 [-6.940 to -0.720] | -1.830 [-4.610 to 0.000]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0118, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0191, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

13. Secondary Outcome: Change in Waist Circumferences
Description: To compare the change in waist circumferences between two groups after 12 weeks of follow-up.
Time Frame: 12 weeks
Population: At V5, Waist circumference data were missing for 12 participants in the GA intervention group (GA) and 8 in the control group, resulting in FAS analysis using 86 GA and 93 control participants. In the PPS group, no data were missing for in GA and in control, so PPS analysis included 79 GA and 91 control participants.
Measure: Median (Inter-Quartile Range); unit: Change in Waist circumferences (cm)
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
Change in Waist circumferences (cm)
  FAS analysis | -4.00 [-7.00 to -1.00] | -2.00 [-5.20 to 0.00]
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -4.00 [-7.00 to -1.00] | -2.00 [-5.50 to 0.00]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; Test type: Superiority; p = 0.0057, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0175, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

14. Secondary Outcome: Percent Change in Waist Circumferences
Description: To compare the rate of change in waist circumferences between the two groups after 12-week of follow-up.
Time Frame: 12 weeks
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent change in waist circumferences
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
Percent change in waist circumferences
  FAS analysis | -4.00 [-7.050 to -1.170] | -2.020 [-5.280 to 0.000]
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -3.960 [-6.600 to -1.120] | -2.170 [-5.360 to 0.000]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; FAS analysis; Test type: Superiority; p = 0.0065, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; PPS analysis; Test type: Superiority; p = 0.0188, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

15. Secondary Outcome: Change in BMI
Description: To compare the change in BMI between two groups after 12 weeks of follow-up.
Time Frame: 12 weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Change in BMI (kg/m^2)
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
Change in BMI (kg/m^2)
  FAS analysis | -0.85 [-1.90 to -0.20] | -0.50 [-1.20 to 0.00]
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -0.80 [-1.90 to -0.20] | -0.50 [-1.20 to 0.00]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; Test type: Superiority; p = 0.0087, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; Test type: Superiority; p = 0.0152, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

16. Secondary Outcome: Percent Change in BMI
Description: To compare the rate of change in BMI between the two groups after 12-week of follow-up.
Time Frame: 12 weeks
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Percent Change in BMI
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
Number analyzed (Participants) | 86 | 93
Percent Change in BMI
  FAS analysis | -3.140 [-6.690 to -0.740] | -1.790 [-4.510 to 0.000]
  PPS analysis: number analyzed (Participants) | 79 | 91
  PPS analysis | -3.000 [-7.090 to -0.740] | -1.820 [-4.560 to 0.000]
Statistical Analysis 1: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; Test type: Superiority; p = 0.0103, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05
Statistical Analysis 2: Comparison: GA guided anti-diabetic therapy adjustment vs current guidelines to adjust treatment; Test type: Superiority; p = 0.0176, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p =0.05

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | GA guided anti-diabetic therapy adjustment | current guidelines to adjust treatment
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/98 | 2/102
Other Adverse Events (participants affected / at risk) | 18/98 | 9/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA guided anti-diabetic therapy adjustment (N=98) | current guidelines to adjust treatment (N=102)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
breast cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GA guided anti-diabetic therapy adjustment (N=98) | current guidelines to adjust treatment (N=102)
hyperuricemia (Metabolism and nutrition disorders) | 10 | 5
dyslipidemia (Metabolism and nutrition disorders) | 4 | 4
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT05227677/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT05227677/SAP_001.pdf